CLINICAL TRIAL: NCT05424237
Title: Efficacy and Feasibility of an eHealth Intervention for Pregnant Women on Diet, Physical Activity and Knowledge Related to Pregnancy
Acronym: EmbarApp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Rubén Martín Payo, Associate professor, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021.490
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 1. Sign consent form and baseline assessments
  2. Usual care
  3. Post intervention assessments
- Interention group (Experimental): 1. Sign consent form and baseline assessments
  2. Usual care + app iNATAL
  3. Post intervention assessments
  Interventions: Behavioral: App intervention

INTERVENTIONS:
Behavioral: App intervention — usual care plus app ussage with the aim of promote healthy behaviors (diet, physical activity and weight)
  Arms: Interention group

SUMMARY:
A pragmatic clinical trial are developed with the aim to assess the effectiveness and feasibility of using an app as complement of the usual care that receive pregnancy women in a sanitary area in the Principado de Asturias (Spain).

Participants are pregnancy women attended in the sanitary area number 3 of the Pincipado de Asturias. As inclusion criteria we will consider: i) aged over 18; ii) pregnant with only 1 fetus; iii) low risk pregnancy; iv) smartphone Access; v) signed the informed consent. As exclusion criteria: i) non-fluent Spanish speaker; ii) do not fill the questionnaires.

A randon sample of 153 women will be recruited consequtively, at the first triemester, from the midwife consulting room. Those women to agreed to participate, and sign the infomred consent, will be anonymizated using a alphanumerical code and asigned (according to a previous randomization distribution by code) to a control or an intervention group.

All women are going to receive the baseline and post intervention questionnaires by email. All women are going to receive the usual care. Adittionally, those in the intervention group, will be prompted to use iNATAL app.

The following questionnaires and measures will be used: uMARS Questionnaire to assess and percentage of app usage tot assess the feasibility; to assess the effectiveness: Motiva.Diaf to assess dietary and physical activity recommendations; ad hoc questionnaire to assess knwoldedge pregnancy related; mother complications during of after the pregnancy period and newborn complications.

The intervention takes all pregnancy period.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18
* pregnant with only 1 fetus
* low risk pregnancy
* smartphone Access
* signed the informed consent

Exclusion Criteria:

* non-fluent Spanish speaker
* do not fill the baseline or post-intervention questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy women
Enrollment: 153 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Following dietary recommendations (mean) | Change from Baseline dietary recommendations at 8 or 9 months (depending the pregnancy)
  For both groups. Compliance with dietary recommendations. We are going to use the Motiva.Diaf questionnaire. It includes 7 questions to assess healthy diatery adherence. Response in dichotomous option 0 (not follow the recommendation) or 1 (follow the recommendation). Total score range from 0 (null dietary compliance) to 7 (best dietary compliance).
Following physical activity recommendations (mean) | Change from Baseline dietary recommendations at 8 or 9 months (depending the pregnancy)
  For both groups. Compliance with dietary recommendations. We are going to use the Motiva.Diaf questionnaire. It includes 5 questions to assess healthy diatery adherence. Response in dichotomous option 0 (not follow the recommendation) or 1 (follow the recommendation). Total score range from 0 (null dietary compliance) to 5 (best dietary compliance).
Change in pregnancy knwoledge (mean) | Change from Baseline dietary recommendations at 8 or 9 months (depending the pregnancy)
  For both groups. Ad hoc questionnaire that includes 10 questions related with pregnancy care. Response in dichotomous option 0 (wrong answer) or 1 (correct answer). Total score range from 0 (null knowledge) to 7 (best knowledge).
App ussage | At the end of the intervention (8-9 after baseline)
  Only for intervention group. Use the app during pregnancy period time. Dichotomous answer (yes or not).
Newborn complications (mean) | From birth to one week after.
  Number of complication suffer by the newborn in the first week after the birth.
Women weigh gain (mean) | From baseline to the end of the intervention (8-9 months after baseline)
  Weigh improvement in kilograms during the pregnancy period time
App quality (mean) | At the end of the intervention (8-9 after baseline)
  Only for intervention group. We are going to use the Spanish version of uMARS to assess the objective and subjetive quality of the app. Both dimensions has a total score range from 1 (lowest quality) to 5 (higher quality).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT05424237/Prot_SAP_000.pdf